CLINICAL TRIAL: NCT06148207
Title: [18F]BF3-BPA Injection for PET Imaging Study of Gliomas in the Brain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, YiHui Guan, Professor, Huashan Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY2023-778
Record Dates: First submitted 2023-11-19; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Cerebral Gliosis; Positron Emission Tomography
MeSH Terms: conditions — Gliosis | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low-dose group (Experimental): Subjects in this group were injected intravenously with 5 ± 1 mCi [18F]BF3-BPA
  Interventions: Radiation: [18F]BF3-BPA Injection for PET Imaging
- High-dose group (Experimental): Subjects in this group were injected intravenously with 9 ± 1 mCi [18F]BF3-BPA
  Interventions: Radiation: [18F]BF3-BPA Injection for PET Imaging

INTERVENTIONS:
Radiation: [18F]BF3-BPA Injection for PET Imaging — Two dosing dose groups were designed, 5±1 mCi or 9±1 mCi, with 20 subjects in each dose group, and the high dose group study was conducted after enrollment in the low dose group was completed.

SUMMARY:
In this clinical study, we proposed to perform [18F]BF3-BPA PET imaging in subjects with gliomas, to observe the binding ability and non-specific binding of the tracer to glioma lesions in vivo, and at the same time to evaluate the effectiveness of [18F]BF3-BPA in the diagnosis and differential diagnosis of glioma, and to evaluate the tolerability and safety of the tracer and the imaging method. The efficacy of [18F]BF3-BPA in the diagnosis and differential diagnosis of gliomas will be evaluated, as well as the tolerability and safety of this tracer and imaging method.

This study will provide a new method for in vivo imaging of gliomas and provide a clear and intuitive imaging basis for clinical diagnosis, differential diagnosis and treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with suspicious brain gliomas:
* Patients diagnosed by the investigator, based on symptoms, course of disease, and MRI of the head, as having a suspected high- or low-grade brain glioma, scheduled for brain tumor resection, and with no contraindications to surgery;
* No prior and/or current surgery, radiotherapy, or puncture biopsy (other than treatment for symptomatic relief) for brain tumors;
* No other primary malignant tumor. 2. age ≥ 18 years; 3. Eastern Cooperative Oncology Group (ECOG) 0-2; 4. adequate organ function:
* Platelet count >100 x 109/L;
* Urea/urea nitrogen and serum creatinine <1.5 times upper limit of normal (ULN);
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times ULN.

  5. Subjects should be fully informed of the content, process and possible risks of the test and voluntarily sign an informed consent form.

Exclusion Criteria:

* Subjects meeting any of the following criteria will be excluded from the study:

  1. Severe allergic reaction to any of the drugs or their components in this trial;
  2. Those who cannot tolerate or are contraindicated to undergo MRI and PET;
  3. Those who cannot accept or tolerate blood sample collection;
  4. Those who are unable to use effective contraception from the date of signing the informed consent to 3 months after the administration of the drug;
  5. pregnant or lactating women or those with positive blood pregnancy test results;
  6. Those who have participated in other interventional clinical trials prior to the date of informed consent and are within 5 half-lives of the trial drug, or are participating in other interventional clinical trials;

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Complete PET imaging | 90mins from time of injection
  To evaluate the biodistribution characteristics (SUVmax, SUVmean) of PET imaging with different doses of [18F]BF3-BPA in brain tumor/normal brain tissues of patients with suspected gliomas, and to obtain the optimal imaging time and optimal dose of [18F]BF3-BPA PET imaging in patients with suspected gliomas.

CONTACTS AND LOCATIONS:
Overall Officials: Fang Xie, PhD, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, China